CLINICAL TRIAL: NCT04576325
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Pharmacokinetic Profile of Voriconazole Inhalation Powder in Adult Subjects With Asthma
Brief Title: Pharmacokinetic Profile of Voriconazole Inhalation Powder in Adult Subjects With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TFF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TFF-V1-002
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: voriconazole; asthmatic; inhaled; VFEND; aspergillosis; IPA; fungal infection; pulmonary aspergillosis
MeSH Terms: conditions — Asthma; Respiratory Aspiration; Aspergillosis; Mycoses; Pulmonary Aspergillosis

STUDY DESIGN:
Intervention Model Description: In each cohort, 8 eligible subjects will be randomized in a 3:1 ratio (6 on active and 2 on placebo) to receive 7 doses (over 3.5 days) of VIP BID or placebo
Who Masked: Participant, Investigator
Masking Description: The investigators, study coordinators, study subjects and the Sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voriconazole Inhalation Powder (Experimental): Investigational drug will be supplied as capsules, each capsule contains 10 mg of Voriconazole Inhalation Powder. The capsules will be administered with the provided breath actuated Plastiape RS00 Model 8 Dry Powder Inhaler device.
  Interventions: Drug: Voriconazole Inhalation Powder
- Placebo (Placebo Comparator): Placebo will be supplied as capsules, each capsule will contain no active ingredient. The capsules will be administered with the provided breath actuated Plastiape RS00 Model 8 Dry Powder Inhaler device.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voriconazole Inhalation Powder — For each dose, multiple inhalations will be required (4 capsules in Cohort 1 and 8 capsules in Cohort 2). All capsules for a given dose must be inhaled over a maximum 10-minute period. Cohort 1 will receive 40 mg BID and Cohort 2 will receive 80 mg BID. Both Cohorts will administer study drug for 3.5 days (7 days total).
  Other Names: VIP
  Arms: Voriconazole Inhalation Powder
Drug: Placebo — For each dose, multiple inhalations will be required (4 capsules in Cohort 1 and 8 capsules in Cohort 2). All capsules must be inhaled over a maximum 10-minute period. Cohort 1 will receive 4 capsules of inactive BID and Cohort 2 will receive 8 capsules of inactive BID. Both Cohorts will administer placebo capsules for 3.5 days (7 days total).
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
This is a Phase 1b, randomized, double-blind, placebo-controlled trial to evaluate the safety, tolerability, and pharmacokinetic profiles of voriconazole inhalation powder in adult subjects with well-controlled asthma. This study will involve 2 cohorts.

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, double-blind, placebo-controlled trial to evaluate the safety, tolerability, and pharmacokinetic (PK) profiles of voriconazole inhalation powder (VIP) in adult subjects with well-controlled Step 2 or Step 3 asthma. This study will involve a minimum of 2 cohorts. The first 2 subjects randomized into each cohort will be sentinel subjects (i.e., one assigned to VIP and one assigned to placebo). If study drug is deemed safe by the PI, the remaining 6 subjects (5 on VIP and 1 on placebo) may be enrolled.

* In Cohort 1, 8 eligible subjects will be randomized in a 3:1 ratio (6 on active and 2 on placebo) to receive 7 doses BID (over 3.5 days) of 40mg VIP or inhaled placebo. Following completion of Cohort 1 and after dose escalation has been approved by the SMC, Cohort 2 may begin.
* In Cohort 2, 8 eligible subjects will be randomized in a 3:1 ratio to receive 7 doses BID (over 3.5 days) of 80 mg VIP or placebo . Doses will be administered twice daily every 12 (± 1 hours).

A third cohort with the same design and number of subjects may be initiated if there are safety or other findings from Cohort 2 that warrant investigation of an intermediary dose (e.g., VIP 60 mg BID). The decision to initiate this potential 3rd cohort will be made by the Sponsor in collaboration with the safety monitoring committee (SMC). A sentinel design will not be required for this cohort.

Following a variable length Screening period, all subjects will be domiciled in a clinical research facility from the Check-In Day (Day -1) and will remain domiciled until the morning of Day 5. A follow-up phone call or clinic visit (depending on best practices at the time for Coronavirus Disease 2019 [COVID-19] precautions) will be made one week later to assess subject status and record any adverse events (AEs).

Safety will be assessed by monitoring AEs, clinical laboratory tests, vital signs, pulse oximetry, spirometry, 12-lead ECGs, and physical examinations. Blood PK will be assessed from serial blood collections following Dose 1 and Dose 7. Study treatment stopping rules for individual subjects will be based on AEs, SAEs, required changes during the treatment period to asthma medications, spirometry measure of forced expiratory volume at 1 second (FEV1), and increases in QTcF values on ECG.

The SMC will review the safety information accrued during the study and will be responsible for reviewing Cohort 1 safety information before authorizing dose escalation to Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to participate and is willing and able to participate in the study and abide by study restrictions in the judgement of the Investigator.
2. Males or non-pregnant, non-lactating females.
3. Well-controlled Step 2 or Step 3 asthma defined by the GINA guidelines.
4. Body mass index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2 at Screening.
5. Normal blood pressure at Screening and Check-In.
6. Normal clinical laboratory tests at Screening and Check-In.
7. Negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody, human immunodeficiency virus (HIV) I and II antibodies, tuberculosis (TB), or COVID-19 at Screening.
8. Able to successfully perform spirometry and use the inhalation device, as demonstrated at Screening and Check-In.

Exclusion Criteria:

1. History or presence of clinically significant medical, ophthalmic, or psychiatric conditions or diseases in the opinion of the Investigator or designee.
2. History or current evidence of any chronic upper or lower respiratory conditions other than asthma or allergic (seasonal or perennial), or non-allergic rhinitis. History of mild acute upper or lower respiratory conditions are allowed, provided that it has been at least 3 months since the condition resolved and provided that in the Investigator's judgement, this occurrence poses no additional risk for this subject.
3. History of any illness or surgery within 6 months of Screening that, in the opinion of the Investigator, might confound the results of the study or that poses an additional risk to the subject by their participation in the study.
4. Current or former smokers, users of e-cigarettes or nicotine replacement products who have more than a 10-pack year history of smoking and who have used these products within the 6 months prior to Screening.
5. History or presence of alcoholism or drug abuse within the past 2 years prior to Screening.
6. History or presence of hypersensitivity or idiosyncratic reaction to voriconazole or any triazole antifungal.
7. Received any marketed or investigational biologic within 4 months or 5 half-lives prior to dosing, whichever is longer.
8. Received treatment with investigational study drug (or device) in another clinical study within 30 days or five half-lives of dosing, whichever is longer.
9. Subjects who have taken any of the protocol prohibited medications within 30 days of the first dose or who are expected to require these medications during the study.
10. ECG with a QTcF interval >450 msec for males or QTcF interval > 470 msec for females or ECG findings deemed clinically significantly abnormal by the Investigator prior to the first dose.
11. Unable to refrain from or anticipates the use of any vitamin supplements, prescription, over-the-counter (OTC), herbal preparations or medications other than those specified for asthma or allergic rhinitis medications, or topical ophthalmic drops beginning 14 days prior to the first dose and throughout the study.
12. Females requiring hormone replacement therapy within 30 days of Screening or during the study.
13. Allergy or sensitivity to lactose or milk products.
14. Donation of blood or blood products within the last 2 months.
15. Loss of 50 to 500 mL whole blood within the past two months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience Adverse Events (AEs), Serious Adverse Events (SAEs) and withdrawals due to AEs | Through study completion, an average of 14 days
  Frequency of AEs, SAEs, and discontinuations due to AEs
Number of participants who experience vital sign abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant vital sign values
Number of participants who experience pulse oximetry abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant pulse oximetry values
Mean change from baseline in forced expiratory volume (FEV1) | Baseline through study completion, an average of 14 days
  Spirometry used to measure FEV1 lung function
Mean change from baseline in forced vital capacity (FVC) | Baseline through study completion, an average of 14 days
  Spirometry used to measure FVC lung function
Mean change from baseline in forced expiratory flow over the middle 1/2 of the FVC (FEF25-75%) | Baseline through study completion, an average of 14 days
  Spirometry used to measure FVC and FEF25-75% lung function
Mean change from baseline in FEV1/FVC ratio | Baseline through study completion, an average of 14 days
  Spirometry used to measure FEV1 and FVC lung function
Mean change from baseline in QTcF changes via ECG | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant ECG values
Number of participants who experience physical examination abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant physical examination findings
Number of participants who experience laboratory test abnormalities | Baseline through study completion, an average of 14 days
  Number of participants with potentially clinically significant laboratory test results

SECONDARY OUTCOMES:
PK of VIP in plasma: Area under the plasma-concentration time curve (AUC) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for plasma analysis
PK of VIP in plasma: Area under the plasma-concentration time curve over the first 12 hours after dosing (AUC0-12) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Area under the concentration time curve, from time 0 to the last observed non-zero concentration (AUC0-tlast) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Area under the concentration time curve from time 0 extrapolated to infinity (AUC∞) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Maximum observed concentration (Cmax) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Time to maximal observed concentration (tmax) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Termination elimination half-life (t½) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Apparent total body clearance (CL/F) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis
PK of VIP in plasma: Apparent volume of distribution during the terminal elimination phase (Vz/F) | Predose Day 1 and through 12 hours post last dose (day 4)
  Blood samples will be collected for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dale Christensen, PhD, Study Director — TFF Pharmaceuticals
Locations (1):
- Q-Pharm Pty Ltd (Nucleus Networks), Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No